CLINICAL TRIAL: NCT03559322
Title: A Prospective, Observational, Post-market Surveillance Study to Evaluate the Long-term Safety and Efficacy of the iNAP® Sleep Therapy System in Adults With Obstructive Sleep Apnea
Brief Title: Real World Experiences of the iNAP® Lite in OSA Adults in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Somnics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: iNAP®-TW-1702
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: iNAP® Lite Sleep Therapy System — Class II intraoral devices for snoring and/or obstructive sleep apnea

SUMMARY:
A Prospective, Observational, Post-market Surveillance Study to Evaluate the Long-term Safety and Efficacy of the iNAP® Lite Sleep Therapy System in Adults with Obstructive Sleep Apnea

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) impacts sleep quality of patients, which contributes significantly to hypertension, stroke, myocardial infarction and other health problems. Intraoral devices, such as tongue retaining devices, palatal lifting devices and mandibular repositioning devices designed to increase the patency of the airway and to decrease airway obstruction, are used to treat OSA. To this end, we are conducting a prospective, observational, post-market surveillance study to evaluate the long-term safety and efficacy of the iNAP® Lite sleep therapy system (iNAP® Lite), a tongue and soft palate retaining intraoral device, in adults with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with OSA with AHI>5

Exclusion Criteria:

* Patients with central sleep apnea (CSA).
* Patients with have severe respiratory disorders such as pulmonary diseases, pneumothorax, etc.
* Patients with loose teeth or advanced periodontal disease.
* Patients with pathologically low blood pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with obstructive sleep apnea in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events in this entire study. | through study completion, up to 10 weeks
  All safety events will be listed and tabulated for their occurrence rate

SECONDARY OUTCOMES:
iNAP® Lite-treated clinical success rate | a treated polysomnography or polygraphy assessment night
  AHI is the number of apnea/hypopnea events divided by total sleep time (TST), i.e., the number of hours of sleep. Clinical success rate is defined as the proportion of patients in the PP cohort with an AHI reduction of >50% and treated AHI <20 on the Tx PSG Study when compared with the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Chu Chen, Ph.D., Study Chair — Somnics, Inc.
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
May or may not share the results in a publication.

REFERENCES:
- [Derived] Lin HY, Nien CT, Chen CC, Hong II, Lin C, Lin CM. Optimizing treatment of the novel intra-oral negative pressure for obstructive sleep apnea. Sleep Breath. 2025 Feb 28;29(1):115. doi: 10.1007/s11325-025-03263-w. PMID 40019614